CLINICAL TRIAL: NCT04484857
Title: Phase 3b Multicenter, Open-Label Single Arm Study of Roxadustat: Either as Conversion From an Erythropoiesis Stimulating Agent (ESA), or as Initial Anemia Treatment in Hemodialysis (HD) Patients
Brief Title: Study of Roxadustat Conversion in Participants Receiving Stable ESA or as Initial Anemia Treatment in Hemodialysis Participants
Acronym: ASPEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-096
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-06

CONDITIONS: Anemia Associated With End Stage Renal Disease
MeSH Terms: interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Roxadustat (Experimental): Participants will receive roxadustat as an oral tablet, 3 times per week (TIW) for up to a maximum of 24 weeks. If a participant require roxadustat <60 milligrams (mg)/week to maintain hemoglobin (Hb) levels, the dose frequency will be reduced in a stepwise manner, for example, to twice weekly (BIW), and then once weekly (QW). For participants converted from an ESA, the initial roxadustat dose will be based on the average prescribed ESA dose in the last 4 weeks (for epoetin alfa and darbepoetin alfa) or 8 weeks (for methoxy polyethylene glycol-epoetin beta [Mircera®]). For participants with <6 weeks of prior ESA use, the initial roxadustat dose will be based on a 2-tiered, weight-based dosing scheme. Dose adjustment evaluations will be made every 4 weeks and doses will be titrated based on Hb level and rate of Hb change. The prescribed dose will not exceed the maximum allowable dose of 3.0 mg/kilogram (kg)/dose or 400 mg per dose, whichever is lower.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be administered per dose and schedule specified in the arm description.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of roxadustat dosing regimens among hemodialysis participants converted from erythropoiesis stimulating agent (ESA) therapy or who are ESA-naïve.

ELIGIBILITY:
Key Inclusion Criteria:

* Receiving chronic dialysis for end stage renal disease (ESRD)
* Vascular access must be a functioning native arteriovenous fistula or graft with adequate flow in the opinion of the investigator, or permanent tunnelled catheter
* Screening Hb criteria: Participants converting from an ESA: between 9.0 to 12.0 grams (g)/deciliter (dL); Participants initiating anemia treatment: < 10.0 g/dL
* Ferritin ≥ 50 nanograms (ng)/mililiter (mL), Transferrin saturation (TSAT) ≥ 10% at screening
* Participant's alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are ≤ 3 x upper limit of normal (ULN), and total bilirubin (TBL) is ≤ 1.5 x ULN at screening and prior to initiating roxadustat treatment.
* Body weight between 45.0 to 160.0 kg

Key Exclusion Criteria:

* Red blood cell (RBC) transfusion within 4 weeks prior to enrollment
* Known history of myelodysplastic syndrome or multiple myeloma
* Known hereditary hematologic disease or other known causes for anemia other than chronic kidney disease (CKD)
* Known chronic inflammatory disease that is determined by the investigator to be the primary cause of anemia
* Active or chronic gastrointestinal bleeding
* Treated with iron-chelating agents within 4 weeks prior to enrollment
* History of New York Heart Association (NYHA) Class III or IV congestive heart failure
* History of myocardial infarction, acute coronary syndrome, stroke, seizure, or a thrombotic/thromboembolic event (excluding vascular dialysis access stenosis/thrombosis) within 12 weeks prior to enrollment
* Uncontrolled hypertension, in the opinion of the Investigator
* Participant has a diagnosis or suspicion (for example, complex kidney cyst of Bosniak Category II or higher) of renal cell carcinoma (Principal Investigator's discretion)
* History of malignancy, except for cancers determined to be cured or in remission for ≥ 2 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Eisner, Study Chair — Kyntra Bio
Locations (23):
- United States (23):
  - Alaska, Anchorage, Alaska
  - Investigator Site, Pine Bluff, Arkansas
  - Investigational Site, Cerritos, California
  - Investigational Site, Victorville, California
  - Investigational Site, Denver, Colorado
  - Investigational Site, Hartford, Connecticut
  - Investigational Site, Coral Gables, Florida
  - Investigational Site, Hollywood, Florida
  - Investigator Site, Dalton, Georgia
  - Investigational Site, Statesboro, Georgia
  - Investigational Site, Roseville, Michigan
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigator Site, Gallup, New Mexico
  - Investigational Site, The Bronx, New York
  - Investigational Site, Austin, Texas
  - Investigator Site, Dallas, Texas
  - Investigational Site, El Paso, Texas
  - Investigational Site, Houston, Texas
  - Investigator Site, San Antonio, Texas
  - Investigational Site, San Antonio, Texas
  - Investigator Sites, San Antonio, Texas
  - Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Roxadustat: Participants received roxadustat as an oral tablet, 3 times per week (TIW) for up to a maximum of 24 weeks. If a participant required roxadustat <60 milligrams (mg)/week to maintain hemoglobin (Hb) levels, the dose frequency was reduced in a stepwise manner, for example, to twice weekly (BIW), and then once weekly (QW). For participants converted from an erythropoiesis stimulating agent (ESA), the initial roxadustat dose was based on the average prescribed ESA dose in the last 4 weeks (for epoetin alfa and darbepoetin alfa) or 8 weeks (for methoxy polyethylene glycol-epoetin beta [Mircera®]). For participants with <6 weeks of prior ESA use, the initial roxadustat dose was based on a 2-tiered, weight-based dosing scheme. Dose adjustment evaluations were made every 4 weeks and doses were titrated based on Hb level and rate of Hb change. The prescribed dose did not exceed the maximum allowable dose of 3.0 mg/kilogram (kg)/dose or 400 mg per dose, whichever was lower.
Period: Overall Study
Arm/Group | Roxadustat
Started | 283
Received at Least 1 Dose of Study Drug | 283
Full Analysis Set (All enrolled participants who provided baseline Hb data and data for at least 1 postbaseline Hb time point.) | 282
Completed | 36
Not Completed | 247
Not completed — Adverse Event | 2
Not completed — Death | 10
Not completed — Withdrawal by Subject | 3
Not completed — Transferred/Relocation | 5
Not completed — Kidney Transplant | 7
Not completed — Other than specified | 4
Not completed — Participants continued an Optional Extension of Roxadustat Treatment | 216

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Roxadustat: Participants received roxadustat as an oral tablet, TIW for up to a maximum of 24 weeks. If a participant required roxadustat <60 mg/week to maintain Hb levels, the dose frequency was reduced in a stepwise manner, for example, to BIW, and then QW. For participants converted from an ESA, the initial roxadustat dose was based on the average prescribed ESA dose in the last 4 weeks (for epoetin alfa and darbepoetin alfa) or 8 weeks (for Mircera®). For participants with <6 weeks of prior ESA use, the initial roxadustat dose was based on a 2-tiered, weight-based dosing scheme. Dose adjustment evaluations were made every 4 weeks and doses were titrated based on Hb level and rate of Hb change. The prescribed dose did not exceed the maximum allowable dose of 3.0 mg/kg/dose or 400 mg per dose, whichever was lower.
Arm/Group | Roxadustat
Number analyzed (Participants) | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91
  Not Hispanic or Latino | 191
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 113
  Race: American Indian or Alaska Native | 17
  Race: Asian | 8
  Race: Native Hawaiian or Other Pacific Islander | 5
  Race: White | 131
  Race: Other | 7
  Race: Not Reported | 2
Baseline Hb [Mean (Standard Deviation); unit: grams (g)/deciliter (dL)] | 10.554 (0.7228)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Mean Hb Value ≥10 g/dL
Description: Percentage of participants with mean Hb value ≥10 g/dL, averaged from Week 16 through Week 24 has been reported. Baseline Hb was defined as the mean of available central laboratory Hb values prior to first dose of study medication including the predose Hb value collected on Day 1. 95% confidence interval (CI) was calculated based on the normal approximation to the binomial distribution.
Time Frame: Week 16 through Week 24
Population: The full analysis set included all enrolled participants who provided baseline Hb data and data for at least 1 postbaseline Hb time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 282
percentage of participants | 83.7 [78.9 to 88.6]

2. Primary Outcome: Mean Hb Change From Baseline to Average Hb From Weeks 16-24
Description: Baseline Hb was defined as the mean of available central laboratory Hb values prior to first dose of study medication including the predose Hb value collected on Day 1. Missing data was imputed using Monte Carlo Markov Chain (MCMC) imputation model.
Time Frame: Baseline, Weeks 16-24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat
Number analyzed (Participants) | 282
g/dL | 0.22 (1.029)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days post last dose of roxadustat (Week 28)
Description: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Arm/Group | Roxadustat
All-Cause Mortality (participants affected / at risk) | 11/283
Serious Adverse Events (participants affected / at risk) | 82/283
Other Adverse Events (participants affected / at risk) | 19/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=283)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 7
Cardiac arrest (Cardiac disorders) | 5
Cardiac failure congestive (Cardiac disorders) | 4
Cardiac failure acute (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Orbital haematoma (Eye disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 2
General physical health deterioration (General disorders) | 1
Organ failure (General disorders) | 1
Treatment noncompliance (General disorders) | 1
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 10
COVID-19 (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Sepsis (Infections and infestations) | 2
Arteriovenous graft site infection (Infections and infestations) | 1
Bone abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Enterobacter sepsis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Arteriovenous graft site pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 1
Fluid overload (Metabolism and nutrition disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremityvvv (Musculoskeletal and connective tissue disorders) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Basal ganglia haemorrhage (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Hydroureter (Renal and urinary disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 5
Hypertensive emergency (Vascular disorders) | 4
Hypertensive urgency (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=283)
COVID-19 (Infections and infestations) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT04484857/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT04484857/SAP_001.pdf